CLINICAL TRIAL: NCT00915668
Title: An Open-Label, Randomized, Crossover Drug-Drug Interaction Study to Assess the Effects of Multiple Doses of JNJ-31001074 on the Pharmacokinetics of a Single Dose of an Oral Contraceptive Containing Ethinyl Estradiol and Levonorgestrel
Brief Title: A Study to Evaluate the Pharmacokinetic Drug Interaction Between Multiple Doses of JNJ-31001074 and a Single Dose of an Oral Contraceptive Containing Ethinyl Estradiol and Levonorgestrel in Women
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial is postponed pending the completion of other ongoing pre-clinical and clinical work.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Clinical Leader Psychiatry, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR016261
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2010-11

CONDITIONS: Pharmacokinetics; Drug Interactions; Healthy
Keywords: Healthy women; Non-childbearing potential; Drug-drug interaction; Oral contraceptive; OC; Ovral-L; ethinyl estradiol; EE; levonorgestrel; JNJ-31001074
MeSH Terms: interventions — bavisant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: JNJ-31001074

SUMMARY:
The main purpose of this research study is to evaluate the effect of multiple doses of an investigational drug known as JNJ-31001074 on the single dose of combination oral contraceptive Ovral-L containing ethinyl estradiol and levonorgestrel in healthy women who cannot bear children. This study will look at the safety, tolerability (how the drug makes you feel) and pharmacokinetics (what your body does to the drug) of either drug alone and in combination in healthy women.

DETAILED DESCRIPTION:
This is an open-label (both the physician and patient know which treatment will be administered), single center randomized, drug-drug interaction study in healthy female volunteers of non-child bearing potential. A total of 32 volunteers will be enrolled. The study consists of a screening phase, an open label treatment period, and end of study/early withdrawal assessments. Volunteers will be randomly assigned to 1 of 2 treatment sequences. The open-label treatment phase will consist of two periods. In each period, volunteers will receive either of the following treatment(s): Treatment A: a single dose of oral contraceptive containing 0.03 mg ethinyl estradiol and 0.15 mg levonorgestrel (Ovral-L) on Day 1 and Treatment B: multiple daily doses of 10 mg JNJ-31001074 on Days 1 to 8 and a single dose of oral contraceptive containing 0.03 mg ethinyl estradiol and 0.15 mg levonorgestrel (Ovral-L) on Day 7. A washout (no treatment break or drug holiday) period of 28 days separates the two occasions of single dose administration of oral contraceptives in Periods 1 and 2. Safety and tolerability will be assessed from the time of informed consent to the end-of-study evaluations or early withdrawal. Volunteers will be instructed to report any serious adverse events that occur up to 30 days following the last dose of study drugs. For Treatment A, the volunteer will receive a single dose of oral contraceptive. For Treatment B, the volunteer will receive 10 mg tablet of JNJ-31001074 once daily orally for eight days (Days 1 to 8) and a single dose of oral contraceptive on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Women of non-child bearing potential (i.e., postmenopausal [no spontaneous menses for at least 2 years] or surgically sterile) 18 to 65 years of age, inclusive
* negative pregnancy test
* body mass index between 18 and 30
* body weight greater than or equal to 50 kilograms

Exclusion Criteria:

* History of or current clinically significant medical illness
* abnormal lab values or physical exams
* pregnant or lactating
* used any hormonal products 3 months before study
* drug or alcohol abuse
* history of smoking or nicotine use, 2 weeks before start of study
* clinically significant allergy
* use of prescription and non-prescription medications within 2 weeks before the start of the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Single-dose pharmacokinetics of a combination oral contraceptive when given in combination with JNJ-31001074. | Blood samples taken over a period of 48 hours after combination treatment

SECONDARY OUTCOMES:
To assess the multiple-dose pharmacokinetics of JNJ-31001074 in female volunteers | over a period of 9 days
To assess the safety and tolerability of multiple doses of JNJ-31001074 while administered alone | over a period of 6 days
To assess the safety and tolerability of multiple doses of JNJ-31001074 while administered together with a single-dose of an oral contraceptive in healthy female volunteers | over a period of 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.